CLINICAL TRIAL: NCT00297921
Title: A Phase 2 Study of Tandutinib in Patients With Newly Diagnosed Acute Myelogenous Leukemia Who Are Considered Ineligible For or Who Decline Treatment With Standard Induction Therapy
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: C03002
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Acute Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — tandutinib

INTERVENTIONS:
Drug: tandutinib

SUMMARY:
Prospective, nonrandomized, noncomparative, open-label, multicenter, 2-stage clinical study designed to determine the overall response (combined complete remission, complete remission with incomplete blood count recovery, partial remission, or blast response) rate following tandutinib therapy in 2 groups of patients with newly diagnosed Acute Myelogenous Luekemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Unequivocal histologic or cytologic diagnosis of AML (based on the WorldHealth Organization [WHO] and/or FAB classifications), excluding acute promyelocytic leukemia (FAB M3).
* AML patients with a history of antecedent MDS or MPD are eligible for treatment in this study.
* In the opinion of the investigator is ineligible for or has declined treatment with standard induction therapy
* ECOG performance status of equal to or less then 3
* Ability to voluntarily provide written informed consent
* Determination of the presence or absence of a FLT3-ITD mutation before enrollment once it is ascertained that determination of FLT3-ITD mutation status is required to avoid exceeding enrollment in either patient group

Exclusion Criteria:

* Presence of an active malignancy other than AML at the time of study entry
* Documented or suspected central nervous system leukemia involvement
* Known gastrointestinal disease that could interfere with the absorption of oral tandutinib
* Severe central nervous system, pulmonary, renal, or hepatic disease not related to AML
* Myocardial infarction within 6 months of enrollment or New York Heart Association (NYHA) Class III or Class IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia or active conduction system abnormalities
* QTc >500 milliseconds (ms)
* Family history of or congenital QTc prolongation
* Pretreatment laboratory test values as follows:

  * Total bilirubin >2.5 x the upper limit of normal (ULN)
  * Alanine aminotransferase (ALT) >2.5 x the ULN
  * Serum creatinine >4.0 mg/dL
* Known or suspected infection with human immunodeficiency virus
* Known active infection with hepatitis B or hepatitis C
* Known or suspected primary muscular or neuromuscular disease (eg, muscular dystrophy or myasthenia gravis)
* Receipt of prior antineoplastic therapy for leukemia, except that prior therapy with the following is allowed:

  * Leukapheresis
  * Treatment for hyperleukocytosis with hydroxyurea
* Receipt of prior antineoplastic therapy for MDS, except that prior therapy with the following is allowed:

  * Growth factor/cytokine support
  * Lenalidomide (Revlimid™)
  * Thalidomide (Thalomid®)
  * Azacitidine (Vidaza®)
  * Decitabine (Dacogen)
* Receipt of prior antineoplastic therapy for MPD, except that prior therapy with the following is allowed:

  * Interferon alpha
  * Anagrelide (Agrylin®)
  * Hydroxyurea
* Antineoplastic, experimental, or radiation therapy within 3 weeks before Day 1, except that hydroxyurea for the treatment of hyperleukocytosis is permitted
* Major surgery within 2 weeks before Day 1
* Men or women of childbearing potential unwilling to use adequate contraception from screening to 30 days after the last dose of tandutinib
* A woman who is pregnant or breast feeding. Confirmation that the patient is not pregnant must be established by a negative serum or urine B-human chorionic gonadotropin (B-hCG) pregnancy test result obtained during the screening period. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)